CLINICAL TRIAL: NCT01653223
Title: A Study of Simvastatin on Myocardial Protection and Cardiac Function Undergoing Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Myocardial Protection Effect of Simvastatin Undergoing Cardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jing-song Ou, Director, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: statin2; 5010-2012001 (Other Grant/Funding Number: Sun Yat-sen University); 5010-2014002 (Other Grant/Funding Number: Sun Yat-sen University)
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Congenital Heart Disease; Heart Valve Disease
MeSH Terms: conditions — Heart Defects, Congenital; Heart Valve Diseases | interventions — Simvastatin; Simcor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control (No Intervention): untreated
- short statin (Experimental): Simvastatin (20 mg) was administered every day for the 5-7 days preoperatively, but not the day of surgery in the statin group. Then simvastatin was re-administered at the second day until 7 days postoperatively.
  Interventions: Drug: simvastatin
- long statin (Experimental): Simvastatin (20 mg) was administered every day for the 5-7 days preoperatively, but not the day of surgery in the statin group. Then simvastatin was re-administered at the second day until 6 months postoperatively.
  Interventions: Drug: simvastatin

INTERVENTIONS:
Drug: simvastatin — In short statin group: 20 mg per day, start at 5-7 days before surgery and continue for 7 days.
  In long statin group: 20 mg per day, start at 5-7 days before surgery and continue for 6 months.
  Other Names: simcor
  Arms: long statin; short statin

SUMMARY:
Statins have been used to low cholesterol to prevent and treat coronary artery diseases. It was also reported that statins could protect endothelial function and cardiac function during coronary artery bypass graft. The investigators recent found simvastatin reduced myocardial injury during noncoronary artery cardiac surgery in single medical center. The investigators further investigate that whether simvastatin can protect myocardium during noncoronary artery cardiac surgery with cardiopulmonary bypass and improve cardiac function with long term use postoperatively in two medical centers.

ELIGIBILITY:
Inclusion Criteria:

* More than 18-year-old,
* Congenital heart disease(not complex),
* Isolated heart valve disease,

Exclusion Criteria:

* Coronary artery disease
* Allergy for statins
* Poor liver function,Hepatitis
* Gestation women and Breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Estimated)
Dates: Start 2013-01; Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
troponin | within the first 7 days after surgery
  The investigator will measure the plasma troponin level in several time points before and after surgery in each patient. This is mainly for the comparason between control and short statin, which has been proved in our previous clinical trial: statin1.
ejection fraction | within two years
  Each patient will be followed up and checked with B ultrasound on heart in 1,3,6,12,18 and 24 months after surgery. The ejection fraction will be measured. This is mainly for the comparason between short statin and long statin, which is the major goal in this clinical trial: statin 2.

SECONDARY OUTCOMES:
long term survival | within two years
  Each patient will be followed up and observed survival time.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-song Ou, MD,PhD, Principal Investigator — The Frist Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Marques Antunes M, Nunes-Ferreira A, Duarte GS, Gouveia E Melo R, Sucena Rodrigues B, Guerra NC, Nobre A, Pinto FJ, Costa J, Caldeira D. Preoperative statin therapy for adults undergoing cardiac surgery. Cochrane Database Syst Rev. 2024 Jul 22;7(7):CD008493. doi: 10.1002/14651858.CD008493.pub5. PMID 39037762